CLINICAL TRIAL: NCT06628232
Title: The Effect of Giving a Pacifier Dipped in Breast Milk, Heel Warming, and Applying Both Together on Pain and Salivary Cortisol Levels During Heel Stick in Preterm Newborns: Randomized Controlled Study.
Brief Title: Effect of Nursing Interventions on Pain and Salivary Cortisol Levels During Heel Stick in Preterm Newborns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Zeynem YILDIRIM BALKAN, Assistant Professor and Principal Investigator, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TNKU-Z.BALKAN-2
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: PreTerm Neonate
Keywords: preterm; leel prick; pain; salivary cortisol; nursing care
MeSH Terms: conditions — Premature Birth; Pain | interventions — Pacifiers; Milk, Human

STUDY DESIGN:
Intervention Model Description: Application of 3 different interventions to reduce pain during heel prick blood collection in newborns and comparison with the control group.
  Control Group 1 (swaddling from mother&amp;amp;#39;s lap) Experiment Group 2 (swaddling from mother&amp;amp;#39;s lap + pacifier) Experiment Group 3 (swaddling from mother&amp;amp;#39;s lap + heel warming) Experiment Group 4 (swaddling from mother&amp;amp;#39;s lap + pacifier + heel warming)
Who Masked: Investigator
Masking Description: The same neonatal nurse with at least 5 years of experience will perform the interventions.
  Salivary cortisol sample will be taken by the same investigator with 5 years of experience.
  Salivary cortisol analysis will be performed in the laboratory by biochemistry specialists who have not seen the interventions performed on the newborn.
  Babies will be video recorded before, during and after the procedure.
  Video recordings will be monitored and recorded by 2 independent investigators.
  Data will be analyzed by an independent statistician other than the researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- pacifier with breast milk group (Experimental): swaddling in the mother's lap together with giving a pacifier dipped in breast milk
  Interventions: Other: pacifier with breast milk
- heel heating group (Experimental): swaddling in the mother's lap together with local dry heat application
  Interventions: Other: heel heating
- combined intervention group (Experimental): all interventions combined (swaddling in the mother's lap together with giving a pacifier dipped in breast milk and heel heating
  Interventions: Other: interventions combined
- Control (Other): swaddling the baby in the mother's lap
  Interventions: Other: Control

INTERVENTIONS:
Other: pacifier with breast milk — swaddling in the mother's lap together with giving a pacifier dipped in breast milk
  Arms: pacifier with breast milk group
Other: heel heating — swaddling in the mother's lap together with local dry heat application
  Arms: heel heating group
Other: interventions combined — swaddling in the mother's lap together with giving a pacifier dipped in breast milk and heel heating
  Arms: combined intervention group
Other: Control — swaddling the baby in the mother's lap
  Arms: Control

SUMMARY:
Babies born before the thirty-seventh gestational week are called preterm or premature. Most preterm newborns require Neonatal Intensive Care Unit (NICU) care depending on their gestational age and clinical condition. Although many painful invasive procedures are usually performed on newborns in the NICU, the most common procedure is heel prick. Heel prick is a painful and stressful procedure for the newborn. Neonates do not respond to pain verbally; they respond physiologically, behaviorally and hormonally. Physiologic responses of preterm infants to pain include increased heart and respiratory rate, increased blood pressure and intracranial pressure, decreased oxygenation, and sweating of palms. Among the hormonal symptoms caused by stress in newborns, the most commonly used biochemical method is the measurement of cortisol level. It is reported that there is a significant correlation between salivary and plasma cortisol levels and salivary cortisol level reflects plasma cortisol level. This method is particularly preferred because saliva sampling is much less stressful.

DETAILED DESCRIPTION:
Health professionals should be able to evaluate pain, reduce or eliminate pain in pain management of neonates in interventional applications. Pharmacologic and nonpharmacologic methods are used in pain management. When these methods are applied together, their effectiveness increases in pain related to invasive interventions. Pharmacologically, opioid analgesics, sedatives and local anesthetics are used. Nonpharmacologic methods include breastfeeding, pacifier, oral sucrose, music, warm application, massage, therapeutic touch and positioning such as nesting, fetal positioning, swaddling, kangaroo care, rocking and holding.

In many studies, nonpharmacologic interventions have been applied and compared to reduce pain during heel prick in preterm newborns. In the routine of the clinic, heel prick blood collection from preterm newborns is performed by hugging the mother in her lap. The swaddling procedure for preterm newborns in the control group is recommended by the American Academy of Pediatrics. The swaddling method supports flexion and lateral posture, which is the developmental position of the newborn. With this position, the newborn comes to its position in the uterus, which is familiar to it, ensuring its physiological stability and improving its capacity. In a systematic review of 3396 participants, preterm newborns were calmed and immediately stabilized by kangaroo care, non-nutritive sucking and swaddling methods. Since these methods reduce pain and stress in preterm newborns, they are also reported to be included in "Individualized Supportive Developmental Care" practices.

Many studies have shown that giving pacifiers to newborns is effective in reducing pain. In addition, oral administration of breast milk alone, without breastfeeding, has been found to reduce pain during heel prick, nasopharyngeal aspiration, venipuncture and retinopathy examination in preterms. In the study conducted by Lan et al., breast milk was sniffed to the newborn during heel prick blood collection or tasted by dropping into the newborns mouth with a syringe. As a result, they reported that sniffing and plus tasting breast milk was effective in alleviating pain in newborns.

In the literature, it is emphasized that the pain that occurs during heel blood collection is closely related to the squeezing of the heel to collect blood, not during the needle insertion into the heel, and it is thought that keeping the newborn in an upright position during heel blood collection may facilitate blood flow through gravity and reduce the amount of squeezing required to obtain the sample. However, there are studies showing that heel warming is effective in reducing pain in newborns. It has been stated that with warm application to the heel -with the effect of vasodilation- fewer needling is performed in the heel, the amount of blood required for the procedure increases and the procedure is completed in a shorter time. It is predicted that the heel of the newborn will be squeezed less thanks to the warm application.

However, there is a very limited number of studies evaluating the effectiveness of different nonpharmacologic interventions during heel prick blood collection and measuring the stress marker cortisol. In addition, no study was found to investigate the effectiveness of other interventions (heel warming and giving a pacifier dipped in breast milk) in combination with wrapping among nonpharmacological interventions.

This study aimed to reduce pain during heel prick blood collection in preterm newborns by swaddling the baby in the mothers lap (control group), swaddling in the mothers lap together with giving a pacifier dipped in breast milk (pacifier with breast milk group), swaddling in the mother;s lap together with local dry heat application (heel heating group), and all interventions combined (swaddling in the mother;s lap together with giving a pacifier dipped in breast milk and heel heating-combined intervention group). In addition, it was planned as a randomized controlled experimental design to determine and compare the effects of these nursing interventions on the newborns physiological parameters, pain, salivary cortisol level, crying and procedure time.

Place and Time to Conduct the Research:

The research will be carried out between November 2024 and August 2025 in the Neonatal Intensive Care Unit of Tekirdag Namik Kemal University Hospital.

Population and Sample of the Study:

The study population will consist of infants who meet the inclusion criteria in the NICU of Tekirdağ Namik Kemal University between 01.11.2024-01.08.2025.

The sample size of the study was determined by power analysis. The study comparing non-nutritive suction, sucrose and combination interventions in heel prick blood collection in newborns with the control group was taken as a basis. According to the PIPP pain assessment scale used in the study, the 1st experimental group had a mean score of 9.3 ± 1.3, the 2nd experimental group 10.1 ± 2, the 3rd group 4.4 ± 1.5, and the control group 13.3 ± 1.6. In this study, it was determined that a total of 88 infants (22 in each group) should be included in the study in the sample number calculation made in the G*Power (3.1.9.2.) program with a 5% alpha margin of error (two-way) and 80% power, predicting that the PIPP score mean difference would have a large effect size (.95 large effect) (the effect size was found to be 2.74).

Randomization:

The sample will be randomly selected from the study population. In the study, randomization of premature newborns will be performed in a computer environment. The newborns to be subjected to heel prick blood collection were placed in groups with a randomized controlled method with 18 babies in each group. In the study, randomization was performed by entering the number of cases through the program whose URL address is http://www.randomizer.org.

Control (swaddling from mothers lap) 76, 41, 70, 15, 43, 38, 63, 2, 28, 55, 30, 35, 86, 61, 57, 84, 80, 74, 3, 24, 83, 71 Experiment 2 (swaddling from mothers lap + pacifier) 18, 79, 23, 19, 48, 47, 2, 61, 10, 73, 35, 74, 87, 38, 32, 5, 11, 12, 49, 80, 44, 55 Experiment 3 (swaddling from mothers lap + heel warming) 25, 17, 50, 7, 64, 35, 45, 11, 48, 82, 73, 23, 32, 54, 49, 74, 79, 3, 68, 56, 24, 81 Experiment 4 (swaddling from mothers lap + pacifier + heel warming) 57, 33, 21, 64, 13, 47, 56, 31, 41, 28, 43, 85, 20, 1, 75, 52, 11, 14, 3, 6, 38, 15

ELIGIBILITY:
Inclusion Criteria:

* Mother 18 years of age or older
* Mother is literate
* Whether the mother gives birth naturally or by caesarean section
* Uncomplicated pregnancy and birth history in mother
* Mother's voluntary participation in the study
* Preterm babies between 34 0/7-36 6/7 weeks
* Prematurity at 34 0/7-36 6/7 weeks and weight appropriate for the week (Appropriate Gestational Age- AGA),
* The baby should be fed at least 1 hour in advance.
* It has been 1 hour since the last painful intervention on the baby.
* 6Heel blood should be taken 6 hours after taking analgesic, sedative and anticonvulsant medications.

Exclusion Criteria:

* The baby has a fever
* The baby receiving oxygen therapy,
* The baby receiving antibiotic treatment
* The baby has a congenital anomaly
* The baby having the bed side and heater underneath
* The baby receiving phototherapy,
* The baby is connected to a mechanical ventilator
* Babies whose blood was not collected on the first attempt

Ages: 34 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac apex beat (HRV) | Through study completion, an average of 1 year.
  HRV will be evaluated before, during and after the heel blood collection. Each baby will be video recorded for 7-10 minutes before, during and after the procedure by the researcher.
Oxygen saturation (SpO2) | Through study completion, an average of 1 year
  SpO2 will be evaluated before, during and after the heel blood collection. Each baby will be video recorded for 7-10 minutes before, during and after the procedure by the researcher. SpO2 will be recorded from this video recording.
Crying time | Through study completion, an average of 1 year
  The baby crying time will be monitored and recorded 5 minutes before the heel prick and 5 minutes during the heel prick
Premature Infant Pain Profile Scale (PIPP-R) | Through study completion, an average of 1 year
  The PIPP-R scale includes 3 behavioral (frowning, squeezing eyes, nasolabial groove), 2 physiological (heart rate and oxygen saturation) and 2 contextual (behavioral state and gestational age) items. In the scoring of the scale, items related to physiological and behavioral items are scored as 0,1,2,3 in each variable, reflecting the difference between baseline and treatment values. Items related to contextual items are scored as 3,2,1,0 before touching the baby. The babys pain is evaluated on a total score. Accordingly, the maximum score for newborns is 21. If the premature infant pain profile is between 0-6 points, the pain level in the infant is mild, between 7-12 points is moderate, and between 13-21 points is severe pain.
  Each baby will be video monitored and recorded for 7-10 minutes before, during and after the procedure. This video recording will be evaluated and recorded according to the Premature Infant Pain Profile Scale.
Salivary cortisol level | Through study completion, an average of 1 year
  Since cortisol shows circadian rhythm in premature infants, samples will be taken at the same time in the morning. Before taking saliva samples, the newborns mouth will be checked and oral care will be given with SF. Saliva samples will be collected with the Salimetrics Salivary Cortisol Kit by holding it in the cheek and sublingual cavity of the newborn for 1-2 minutes. The samples will be sent to the biochemistry laboratory of the research hospital. The samples will be analyzed for quantitative determination of cortisol by 2 biochemistry experts using standard procedures in the Biochemistry laboratory of TNKU Hospital.
  Samples will be taken twice, both during the procedure and 25 minutes after the procedure (the highest cortisol level after pain in newborns is detected between 20-30 minutes after the procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Zeynem YILDIRIM BALKAN, Assist.Prof., Study Director — Namik Kemal University; Birsen Mutlu, Assoc.Prof., Principal Investigator — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shu SH, Lee YL, Hayter M, Wang RH. Efficacy of swaddling and heel warming on pain response to heel stick in neonates: a randomised control trial. J Clin Nurs. 2014 Nov;23(21-22):3107-14. doi: 10.1111/jocn.12549. Epub 2014 Jan 30. PMID 24476226
- [Result] Badiee Z, Nassiri Z, Armanian A. Cobedding of twin premature infants: calming effects on pain responses. Pediatr Neonatol. 2014 Aug;55(4):262-8. doi: 10.1016/j.pedneo.2013.11.008. Epub 2014 Mar 30. PMID 24694748